#### Protocol KAN-101-03

# A PHASE 2A DOUBLE-BLIND, PLACEBO-CONTROLLED, STUDY TO EVALUATE THE EFFICACY, SAFETY, AND TOLERABILITY OF KAN-101 IN PARTICIPANTS WITH CELIAC DISEASE

Statistical Analysis Plan (SAP)

Version: 6

**Date:** 03Feb2025

# TABLE OF CONTENTS

| LIST OF TABLES | 4 |
|------------------------------------------------------------------|----|
| LIST OF FIGURES | 4 |
| APPENDICES | 4 |
| 1. INTRODUCTION | 9 |
| 1.1. Study Objectives, Endpoints, and Estimands | 9 |
| 1.1.1. Primary Estimand | 10 |
| 1.1.2. Secondary Estimand | 10 |
| 1.2. Study Design | 11 |
| 1.3. Sample Size | 11 |
| 2. ENDPOINTS AND BASELINE VARIABLES: DEFINITIONS AND CONVENTIONS | 12 |
| 2.1. Primary Endpoint | 12 |
| 2.2. Secondary Endpoints | 12 |
| 2.3. Exploratory Endpoints | 13 |
| 2.4. Demographic and Baseline Variables | 15 |
| 2.5. Safety Endpoints | 15 |
| 2.5.1. Adverse Events | 15 |
| 2.5.2. Safety Laboratory Data | 16 |
| 2.5.3. Vital Signs | 17 |
| 3. ANALYSIS SETS | 17 |
| 4. GENERAL METHODOLOGY AND CONVENTIONS | 18 |
| 4.1. Hypotheses and Decision Rules | 18 |
| 4.2. General Methods | 18 |
| 4.2.1. Analyses for Continuous Endpoints | 18 |
| 4.3. Methods to Manage Missing Data | 19 |
| 5. ANALYSES AND SUMMARIES | 19 |
| 5.1. Primary Endpoint Analysis: Vh:Cd | 19 |
| 5.1.1. Main Analysis | 20 |
| 5.1.2. Sensitivity/Supplementary Analysis | 20 |
| 5.2. Secondary Endpoints | 20 |
| 5.2.1. GC IL-2 | 20 |

| 5.2.1.1. Main Analysis | 20 |
|-----------------------------------------------------------------|----|
| 5.2.1.2. Sensitivity/Supplementary Analysis | 20 |
| 5.2.2. IEL density in duodenum biopsy | 20 |
| 5.2.2.1. Main Analysis | 20 |
| 5.2.2.2. Sensitivity/Supplementary Analysis | 20 |
| 5.2.3. Incidence and Severity of TEAEs as Assessed by the CTCAE | 21 |
| 5.2.4. Incidence of Development of ADA During the Study | 21 |
| 5.2.5. PK Concentration. | 21 |
| 5.2.6. PK Parameters | 21 |
| 5.3. Tertiary/Exploratory | 21 |
| 5.3.1. Change from baseline in Marsh-Oberhuber score at Day 29 | 21 |
| 5.3.2. CDSD | 21 |
| 5.3.2.1. PGIS | 22 |
| 5.3.2.2. PGIC | 22 |
| 5.3.2.3. Subset Analyses | 23 |
| 5.4. Baseline and Other Summaries and Analyses | 23 |
| 5.4.1. Baseline Summaries | 23 |
| 5.4.2. Study Conduct and Subject Disposition | 23 |
| 5.4.3. Study Treatment Exposure | 23 |
| 5.4.4. Gluten Challenge | 23 |
| 5.4.5. Concomitant Medications and Non-Drug Treatments | 23 |
| 5.5. Safety Summaries and Analyses | 23 |
| 5.5.1. Adverse Events | 24 |
| 5.5.2. Safety Laboratory Data | 24 |
| 5.5.3. Vital Signs | 24 |
| 6. INTERIM ANALYSES | 24 |
| 7. CHANGES FROM PROTOCOL | 24 |
| 8. REFERENCES | 25 |

# LIST OF TABLES

| Table 1 Summary of Changes | 5 |
|---|---|
| Table 2 Objectives, Endpoints, and Estimands | 9 |
| Table 3 Analysis Windows for PGIS and PGIC | 29 |
| Table 4 Analysis Windows for Vital Signs | 29 |
| Table 5 Analysis Windows for Laboratory Tests | 30 |
| Table 6 Analysis Windows for ADA | 30 |
| Table 7 Analysis Windows for biopsy endpoints (Vh:Cd ratio, IEL density, Marsh-Oberhuber score) | 30 |
| Table 8 Analysis Windows for IL-2 and CDSD at Day 15 (first GC Day) | 30 |
| LIST OF FIGURES Figure 1 Study Design Schema APPENDICES | 11 |
| Appendix 1. Summary of Efficacy/Exploratory Analyses | 26 |
| Appendix 2. Data Derivation Details | 29 |
| Appendix 2.1. Definition and Use of Analysis Windows in Reporting | 29 |
| Appendix 2.2. Celiac Disease Symptom Diary (CDSD) | 31 |
| Appendix 2.3. Patient Global Impression of Severity (PGIS) | 32 |
| Appendix 2.4. Patient Global Impression of Change (PGIC) | 32 |
| Appendix 3. List of Abbreviations. | 33 |

# **VERSION HISTORY**

This Statistical Analysis Plan (SAP) for study KAN-101-03 is based on the protocol Amendment 1 dated 20Mar2024.

**Table 1 Summary of Changes** 

| Version/Date | Associated<br>Protocol<br>Amendment | Rationale | Specific Changes |
|---|---|---|---|
| 1 | Original | Not Applicable (N/A) | N/A |
| 06Nov2023 | 06Sep2023 | | |
| 2<br>05Apr2024 | Amendment 1 20Mar2024 | The protocol was amended based on PART 1 questions received from the EU CTA, submitted 27 Nov 2023 To address FDA comments, received in November 2023 | Section 6, Interim Analyses (IA) updated to provide rationale for having the IA. Section 3, mITT population was added for supplementary analysis purpose. Section 5 and Appendix I, added supplementary analysis for the primary and secondary efficacy endpoints using all collected data (ie, treatment policy) for FAS. Section 5 and Appendix I, added supplementary analysis for the secondary/exploratory efficacy endpoints using all collected data for mITT. |
| | | | Appendix 2, added analysis visit window for ADA. |

**Table 1 Summary of Changes** 

| Version/Date | Associated<br>Protocol<br>Amendment | Rationale | Specific Changes |
|---|---|---|---|
| 3<br>07Jun2024 | Amendment 1 20Mar2024 | Update Section 6 interim analyses | Added sample size calculation and alpha spending for interim analysis in the design section. Changed "intercurrent events" to be included in the population definition. Eliminated the mITT population and replaced with SAS (ITT) population as a sensitivity analysis. Included a BAS |
| 4<br>16Oct2024 | Amendment 1 20Mar2024 | Update Appendix 2.1 | (Biopsy Analysis Set). Analysis windows were updated. |
| | | Added summary and analysis for Nausea Score and Vomiting Frequency and change from baseline | Sections 2.3 and 5.3.2, CDSD 1-Day, 3-Day, 7-Day Nausea Score and Vomiting Frequency and change from baseline at each timepoint post-gluten challenge will be summarized and analyzed using Wilcoxon Signedrank test for within treatment paired comparison and Wilcoxon Rank Sum test for comparison between placebo vs each of KAN group. |
| 5<br>13Dec2024 | Amendment 1 20Mar2024 | Made clarification for CDSD average calculation. | Section 2.3, 5.3.2,<br>Appendix 2.2, CDSD<br>average score calculation<br>was updated.<br>Intent-To-Treta (ITT) was |
| | | Made clarification for analysis set. | removed from Sections 3, 5.1.2, 5.2.2. |

**Table 1 Summary of Changes** 

| Version/Date | Associated<br>Protocol<br>Amendment | Rationale | Specific Changes |
|---|---|---|---|
| | | Marsh-Oberhuber score is categorical | Section 5.3.1, Baseline and Day 29 Marsh-Oberhuber score will be summarized with frequency and percentage. Change from baseline to Day 29 will be summarized using shift table |
| | | COVID-19 pandemic is over. | Section 5.5, COVID-19 listing and summary were removed |
| | | Map IL-2 and CDSD data to Day 15 if first GC is on Day 14 or Day 16. | Appendix 2.1, Analysis window for IL-2 and CDSD was added (Table 8) |
| 03Feb2025 | Amendment 1 20Mar2024 | How to handle CDSD multiple records on a same day | Section 5.3.2, added a statement: If there are multiple records on a same day, the earliest one will be used for analysis. |
| | | Make GC start day window wider | Section 5.3.2, added weekly time definition of analysis window for Week 2 and Week 3 when the first GC day is at Day 17. |
| | | | Appendix Table 8,<br>analysis window for first<br>GC day was changed from<br>"Day 14 to Day 16" to<br>"Day 14 to Day 17". |

**Table 1 Summary of Changes** 

| Version/Date | Associated<br>Protocol<br>Amendment | Rationale | Specific Changes |
|---|---|---|---|
| | | Updated analysis windows for PGIS, PGIC, vital signs, and lab tests. | Appendix 2 Tables 3, 4, 5: analysis windows of Day 15 and Day 29 were updated to relative to the first (or second) GC day instead of absolute study day. |

#### 1. INTRODUCTION

Study KAN-101-03 is a multi-center, double-blind, placebo-controlled Phase 2a study to examine whether KAN-101 confers protection from gluten challenge (GC)-induced histological changes in the duodenum and to further evaluate the safety/tolerability of KAN-101 in adult patients (≥18 years) with celiac disease (CeD).

This SAP provides the detailed methodology for summary and statistical analyses of the data collected in study KAN-101-03. This document may modify the plans outlined in the protocol; however, any major modifications of the primary endpoint definition or its analysis will also be reflected in a protocol amendment.

#### 1.1. Study Objectives, Endpoints, and Estimands

Study objectives, corresponding endpoints, and estimands are provided in the Table 2 below.

Table 2 Objectives, Endpoints, and Estimands

| Objectives | Endpoints | Estimands |
|---|---|---|
| Primary: | Primary: | Primary: |
| Assess the ability of KAN-101 to attenuate GC-induced changes in duodenal histology as measured by changes in villus-height:crypt depth (Vh:Cd) ratio after a 2-week GC. | Changes from baseline in Vh:Cd ratio as assessed by esophagogastroduodenoscopy (EGD) with biopsy after 2-week GC (at Day 29). | Estimand 1: a hypothetical estimand (Section 1.1.1). |
| Secondary: | Secondary: | Secondary: |
| Examine the impact of KAN-101 on biomarker response (interleukin-2 [IL-2]) in peripheral blood following GC | IL-2 change from Day 15 (first day of GC) pre GC to Day 15 post GC. | Estimand 2: a hypothetical estimand (Section 1.1.2). |
| Determine the effects of KAN-101 on histologic features (intraepithelial lymphocytes [IELs] density) in duodenum biopsies following 2-week GC. | Changes from baseline in IEL density in duodenum biopsy after 2-week GC (at Day 29) | Estimand 3: a hypothetical estimand (Section 1.1.2). |
| Assess the safety and tolerability of KAN-101 in participants with CeD. | Incidence and severity of treatment emergent adverse events (TEAEs) as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v6.0 (or higher). | Not applicable. |
| | Incidence and titer of KAN-101 anti-drug antibodies (ADA). | Not applicable. |
| Assess the pharmacokinetics (PK) of multiple doses of KAN-101 in participants with CeD. | Plasma concentration of KAN-101, and associated KAN-101 parameters: AUC <sub>inf</sub> , AUC <sub>last</sub> , C <sub>max</sub> , T <sub>max</sub> and t <sub>½</sub> | Not applicable. |

Table 2 Objectives, Endpoints, and Estimands

| Objectives | Endpoints | Estimands |
|---|---|---|
| Tertiary/Exploratory: | Tertiary/Exploratory: | Tertiary/Exploratory: |
| Evaluate changes in histological features (Marsh-Oberhuber score) after 2-week GC | Changes from baseline in Marsh-Oberhuber score after 2-week GC (at Day 29) | Not applicable. |
| Assess the impact of KAN-101 administration on the incidence of CeD symptoms before and during GC as measured using CDSD v2.1. | Changes from baseline in symptoms PROs including: CDSD v2.1, PGIC and PGIS over time. | Not applicable. |
| Assess whether KAN-101 affects the incidence and/or titer of post-GC celiac serology. | Change from baseline in incidence and titer of tTG IgA and DGP IgG at Day 42. | Not applicable. |

#### 1.1.1. Primary Estimand

Estimand 1: The primary estimand is the hypothetical estimand, which estimates the treatment effect of KAN-101 vs placebo (PBO) for change from baseline in Vh:Cd ratio. It includes the following 5 attributes:

- Population: Participants who receive all 3 doses of study intervention and complete at least 7 days of GC and do not receive prohibited medications.
- Variable: Vh:Cd ratio change from baseline at Day 29.
- Treatment conditions: KAN-101 or PBO.
- Intercurrent Events: Events are addressed in the analysis set definition.
- Population level summary: The least-squares mean (LSM) difference of the change from baseline in Vh:Cd ratio between KAN-101 and PBO.

#### 1.1.2. Secondary Estimand

Estimand 2 is the hypothetical estimand, which estimates the treatment effect of KAN-101 vs PBO for IL-2. It includes the following 5 attributes:

- Population: Participants who receive all 3 doses of study intervention, complete GC at Day 15 and do not receive prohibited medications.
- Variable: log transformed IL-2 change from pre GC to post GC at Day 15.
- Treatment condition: KAN-101 or PBO.
- Intercurrent Events: Events are addressed in the analysis set definition.

• Population level summary: The LSM difference of the change from pre GC to post GC at Day 15 (log transformed) between KAN-101 and PBO.

Estimand 3 is the hypothetical estimand, which estimates the treatment effect of KAN-101 vs PBO for change from baseline in duodenal IEL density. It includes the following 5 attributes:

- Population: Participants who receive all 3 doses of study intervention and complete at least 7 days of the 2-week GC and do not receive prohibited medications.
- Variable: IEL change from baseline at Day 29.
- Treatment conditions: KAN-101 or PBO.
- Intercurrent Events: Events are addressed in the analysis set definition.
- Population level summary: The LSM difference of the change from baseline in IEL between KAN101 and PBO.

#### 1.2. Study Design

Study KAN-101-03 is a multi-center, double-blind, PBO-controlled Phase 2a study to examine whether KAN-101 confers protection from GC-induced histological changes in the duodenum and to further evaluate the safety/tolerability of KAN-101 in adult patients (≥18 years) with CeD. Approximately fifty-two patients (26 patients per arm) will be randomized 1:1 to 0.6 mg/kg KAN-101 (Arm 1) or PBO (Arm 2).

Figure 1 Study Design Schema



#### 1.3. Sample Size

A sufficient number of participants will be screened to achieve approximately 52 treated participants (26 per study arm). The sample size calculation is based on the primary efficacy estimand and its endpoint, changes from baseline in the ratio of Vh:Cd at Day 29 visit. With

an overall 2-sided type I error rate of 5%, the study will have approximately 94% power under a sample size of 26 participants per arm to detect a treatment difference in LSM of 0.50 in change in ratio of Vh:Cd between treatment arms, assuming that the common standard deviation is 0.5 and the difference between the means is 0.5. To adjust for multiple looks, the O'Brien-Fleming adjustment is applied to control overall type I error rate to ensure that the overall Type I error rate remains at 5%. The interim analysis will be evaluated at significance level 0.003 and the final look will be evaluated at significance level 0.049.

# 2. ENDPOINTS AND BASELINE VARIABLES: DEFINITIONS AND CONVENTIONS

#### 2.1. Primary Endpoint

• Change from baseline in Vh:Cd ratio as assessed by EGD with biopsy after 2-week GC (at Day 29).

The biopsy will be performed at screening and Day 29, or ET visit. The Baseline is the last non-missing Vh:Cd ratio at screening.

#### 2.2. Secondary Endpoints

- GC IL-2 change from Day 15 (first day of GC) pre-GC to Day 15 post GC.
  - GC IL-2 will be log transformed prior to calculating the change.
- Change from baseline in IEL density in duodenum biopsy after 2-week GC (at Day 29).

The biopsy will be performed at screening and Day 29, or ET visit. The Baseline is the last non-missing IEL density at screening.

• Incidence and severity of TEAEs as assessed by the CTCAE.

See Section 2.5.1.

• Incidence and titer of KAN-101 ADA.

Positive of ADA will be assessed at Days 1, 7, 29, 42 or early termination (ET) visit.

• Plasma concentration of KAN-101, and associated KAN-101 parameters: AUC<sub>inf</sub>, AUC<sub>last</sub>,  $C_{max}$ ,  $T_{max}$  and  $t_{1/2}$ .

| Parameter | Definition | Method of Determination |
|---|---|---|
| AUC <sub>last</sub> | Area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (C <sub>last</sub> ) | Linear/Log trapezoidal method |
| AUCinf | Area under the plasma concentration-time profile from time 0 extrapolated to infinite time | AUC <sub>last</sub> + (C <sub>last</sub> /K <sub>el</sub> ), where Clast is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis |
| $C_{max}$ | Maximum plasma concentration | Observed directly from data |
| $T_{max}$ | Time to first occurrence of C <sub>max</sub> | Observed directly from data. |
| t <sub>1/2</sub> a | Terminal elimination half-life | Log <sub>e</sub> (2)/K <sub>el</sub> , where K <sub>el</sub> is the terminal Phase rate constant calculated by a linear regression of the loglinear - concentration time- curve. Only those data points judged to describe the terminal log-linear decline will be used in the regression |

• a. If data permits.

# 2.3. Exploratory Endpoints

- Changes from baseline in Marsh-Oberhuber score assessed via EGD with biopsy after 2-week GC.
- The biopsy will be performed at screening and Day 29, or ET visit. Baseline is the last non-missing Marsh-Oberhuber score at screening.
- CDSD

- CDSD is a patient reported outcome (PRO) questionnaire collected daily. The version 2.1 includes 5 severity items and 3 frequency supplement questions (see Appendix 2.2) that will be collected daily.
  - CDSD Total Score is the sum of all 5 severity items. The CDSD Weekly Average Total Score will be calculated, for details on the calculation see below, Section 5.3.2 and Appendix 2.2.
  - The CDSD Gastrointestinal (GI) Domain Score is the sum of items 1-4. The CDSD Weekly Average Gastrointestinal (GI) Domain Score will be calculated, for details on the calculation see below, Section 5.3.2 and Appendix 2.2.
  - For CDSD Nausea score and vomiting frequency, in addition to weekly average score, 3-day average will be derived as well (every 3 days start from Day 15 GC until Day 41). If 2 observations are missing, the 3-day average score will not be calculated. Day 15 Nausea score and vomiting frequency will be analyzed as well.
- For CDSD Total score, GI Domain score, individual severity item and frequency supplement question, the Baseline value is the average of most recent 7-day interval scores before Day 1 (not include Day 1) with at least 4 days with non-missing scores, and will be used as the baseline to calculate the change from baseline to the 1-day, 3-day average and weekly average. If there are ≥4 days missing scores in any 7-day interval before Day 1, the baseline value is set as missing.
- For post-baseline weekly average score calculation, Week 1 is from Day 1 to Day 7, Week 2 is from Day 8 to the day before Day 15 GC, Week 3 is from the day after Day 15 GC to Day 21. The number of days for Week 2 and Week 3 maybe equal to, less than, or greater than 7. See Section 5.3.2 for the details. The weekly average score is the weekly sum score divided by the number of days with non-missing in that week. If daily scores are missing for more than half of total days in a specific week, the average score is missing for that week.
- Change from baseline at each timepoint = observed (or derived as described above) value at each timepoint baseline.
- The observed value and the change in PGIS
- PGIS is a PRO questionnaire designed to assess the patient's impression of disease severity over the past week (see Appendix 2.3) that is collected at baseline (Day 1), Day 15, 29, 42, or ET visit.
- Change from baseline at each timepoint = observed value at each timepoint baseline. Baseline is the last non-missing value up to Day 1.
- The observed value in PGIC

- PGIC is a PRO questionnaire designed to assess the patient's impression of the overall change in participant's celiac disease since receiving study intervention (see Appendix 2.4) that will be collected at Days 15, 29, 42, or ET visit.
- Change from baseline in incidence and titer of tTG IgA and DGP IgG at Day 42.
- Other exploratory biomarkers may be analyzed at a later date.

#### 2.4. Demographic and Baseline Variables

Demographic and baseline characteristics include:

- Age
- Sex
- Race
- Ethnicity
- Height (in cm)
- Weight (in kg)
- Body Mass Index
- Duration of CeD
- Duration of gluten-free diet (GFD)
- CeD Serology at diagnosis
- Histology at diagnosis

#### 2.5. Safety Endpoints

Safety will be assessed by medical history, vital signs, clinical laboratory tests, and the reporting of AEs, in all participants who received any portion of study intervention. Unscheduled safety assessments may be performed at any time during the study to assess any perceived safety concerns. Investigators and Clinicians will review individual participant data throughout the conduct of the study to ensure participants' wellbeing.

#### 2.5.1. Adverse Events

Incidence and severity of TEAEs is the Secondary endpoint.

An adverse event (AE) is considered TEAE to a given treatment if the event start date is on or after the treatment period start date and before end of study.

The CTCAE displays Grades 1 through Grade 5 with unique clinical descriptions of severity for each AE based on below general guideline:

- o **Grade 1:** Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
- o **Grade 2:** Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental activities of daily living (ADL).
- Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting selfcare ADL.
- o **Grade 4:** Life-threatening consequences; urgent intervention indicated.
- Grade 5: Death related to AE.

#### 2.5.2. Safety Laboratory Data

Safety laboratory testing will be performed at Screening, Days 1, 4, 7, 15, 29, 42, or ET visit. The details are listed in below table.

| Hematology | Chemistry | Urinalysis | Other |
|---|---|---|---|
| Hemoglobin | Urea and creatinine | Local | At screening: |
| Hematocrit | Serum cystatin C | dipstick: | FSH <sup>b</sup> |
| RBC count | eGFR | pН | Pregnancy test (β-hCG) <sup>c</sup> |
| Platelet count | Glucose (fasting) | Glucose | HBsAg and HBcAb. |
| WBC count | Calcium | (qual) | HBsAb and HBV |
| Total neutrophils (Abs, %) | Sodium | Protein | DNA as reflex tests |
| Eosinophils (Abs,%) | Potassium | (qual) | Hepatitis C antibody and HCV |
| Monocytes (Abs,%) | Chloride | Blood | RNA as reflex test |
| Basophils (Abs,%) | Total CO <sub>2</sub> (bicarbonate) | (qual) | HIV |
| Lymphocytes (Abs,%) | AST, ALT | Ketones | HLA genotype and CeD |
| PT | Total and direct bilirubin | Nitrites | serology (eg, HLA DQ2.5 and |
| aPTT | Alkaline phosphatase | Leukocyte | HLA-DQ8 testing <sup>d</sup> , |
| INR | Uric acid | esterase | tTG and DGP IgA/IgG) |
| | Albumin | <u>Laboratory:</u> | |
| | Total protein | Microscopy | Biomarker: IL-2 |
| | Magnesium | and culturea | |
| | Amylase | | PK/ADA |
| | Lipase | | |
| | Phosphorus | | |

- a. Only if Urinary Tract Infection is suspected and urine dipstick is positive for nitrites or leukocyte esterase or both.
- b. For confirmation of postmenopausal status only.
- c. A serum pregnancy test is required at screening. Following screening, local urine testing will be standard for the protocol unless serum testing is required by local regulation or IRB/EC. Serum or urine β-hCG for female participants of childbearing potential.
- d. For re-screening, the HLA does not need to be repeated and CeD serology (the tTG and DGP antibody tests) should only be repeated if >3 months have elapsed from end assessment.

#### 2.5.3. Vital Signs

Vital signs will be assessed at Screening, Days 1, 4, 7, 15, 29, 42, or ET visit.

### 3. ANALYSIS SETS

For purposes of analysis, the following analysis sets are defined:

| Analysis Set | Description |
|---|---|
| Enrolled | All participants who sign the ICD. |
| Biomarker Analysis | All participants who are randomly assigned to study |
| Set (BAS) | intervention, receive any portion of study intervention, and |
| | have completed the GC on Day 15, without prohibited |
| | medications. |
| | Participants will be analyzed according to the intervention they |
| | are randomized. |
| Full analysis set | All participants who are randomly assigned to study |
| (FAS) | intervention, receive all 3 doses of study intervention, and |
| | complete at least 7 days of the 2-week GC without prohibited |
| | medications. Participants will be analyzed according to the |
| | intervention they are randomized. |

| Analysis Set | Description |
|---|---|
| Per protocol set | The PPS will include all participants from the FAS who |
| (PPS) | complete all 14 days of the 2-week GC and biopsies, and |
| | without major protocol violations that might affect the |
| | evaluation of the effect of study intervention on the primary |
| | endpoint. The PPS will be used in sensitivity analyses of the |
| | primary and secondary endpoints. Specific reasons for |
| | warranting exclusion from this population will be |
| | documented prior to database lock. |
| Safety analysis set | All participants who receive any portion of study |
| (SAS) | intervention. Participants will be analyzed according to the |
| | intervention they actually received. |
| PK analysis set | All participants who receive any portion of study |
| (PKAS) | intervention and have at least one concentration value. |

#### 4. GENERAL METHODOLOGY AND CONVENTIONS

#### 4.1. Hypotheses and Decision Rules

This protocol is designed to establish the superiority of KAN-101 to PBO for the primary endpoint of the change in Vh:Cd ratio at Day 29. The null hypothesis is that there is no difference between KAN-101 and PBO, and the alternative hypothesis is that there is a significant difference between KAN-101 and PBO. KAN-101 will be considered superior to PBO with the change in Vh:Cd ratio at Day 29, at the interim look, if the difference is statistically significant at the 2-sided 0.003 level. Even if significance is reached at the interim analysis, no decision to stop the trial will be made unless a safety concern arises. Statistical significance will be evaluated at the end of study at the 2-sided 0.049 level.

#### 4.2. General Methods

In general, count and percent will be presented for categorical variables. Number of observations, mean, standard deviation (SD), minimum (min), 1<sup>st</sup>, 2<sup>nd</sup>, 3<sup>rd</sup> quartiles, and maximum (max) will be presented for continuous variables. The coefficient of variation (CV, defined as SD/Mean; %CV=100\*CV), geometric mean (GM), and geometric mean ratio (GMR) will also be included, where appropriate. Graphics will be used to present the data.

#### 4.2.1. Analyses for Continuous Endpoints

For continuous endpoints, the change from baseline will be analyzed by timepoint using analysis of covariance (ANCOVA) model with treatment as a factor, baseline as a covariate. For endpoints without baseline, analysis of variance (ANOVA) model with treatment as a factor will be used for the analysis. Comparison of KAN-101 to PBO (providing LSM of the treatments, LSM of the treatment difference, p-value and 95% CI) will be generated.

#### 4.3. Methods to Manage Missing Data

If a PK concentration value is below Lower Limit of Quantification (LLOQ), that concentration value will be treated as 0 for all analysis. For IL-2, values below LLOQ will be treated as ½LLOQ. Other missing values will not be imputed for safety, efficacy and PK endpoints.

#### 5. ANALYSES AND SUMMARIES

In general, observed values and change from baseline (where applicable) will be descriptively summarized by treatment group with number of observations, mean, SD, min, 1<sup>st</sup>, 2<sup>nd</sup> (median) and 3<sup>rd</sup> quartiles, and max, unless otherwise specified. For log-transformed values the geometric mean and 95% CI will be presented with the summary statistics.

Data will be summarized and analyzed by treatment group for the main population of interest and a separate sensitivity/supplementary analysis(ses) based on the chosen analysis set from Section 3).

| Endpoint | Analysis Set Applied for<br>Main Analysis | Analysis Set Applied for<br>Sensitivity/Supplementary<br>Analysis |
|---|---|---|
| Biopsy (Vh:Cd, IEL Density<br>Marsh-Oberhuber Score) | Full Analysis Set | Per Protocol Set and Safety<br>Analysis Set |
| Biomarker (IL2) | Biomarker Analysis Set | Per Protocol Set and Safety<br>Analysis Set |
| PK | PK Analysis Set | N/A |
| PRO (CDSD, PGIS, PGIC) | Full Analysis Set | N/A |
| Demography and Safety | Safety Analysis Set | N/A |
| ADA | Safety Analysis Set | N/A |

#### 5.1. Primary Endpoint Analysis: Vh:Cd

The primary endpoint is the change from baseline in Vh:Cd ratio as assessed by EGD with biopsy after 2-week GC (at Day 29).

Raw data will be descriptively summarized by treatment group with number of observations, mean, SD, min, 1<sup>st</sup>, 2<sup>nd</sup> and 3<sup>rd</sup> quartiles, and max for the FAS.

#### 5.1.1. Main Analysis

The Hypothetical estimand, Estimand 1 (Section 1.1.1) will be addressed with the following analysis: change from baseline in Vh:Cd ratio at Day 29 will be analyzed using ANCOVA model (Section 4.2.1) for the FAS Population. The LSM change from baseline and associated 95% CI, LSM difference of the change from baseline between KAN-101 and PBO, 95% CI, and p-value will be presented along with summary statistics.

# 5.1.2. Sensitivity/Supplementary Analysis

Per-protocol (PP) additional sensitivity/supplementary analyses will be performed for change from baseline in Vh:Cd ratio at Day 29 visit using the same approach of main analysis as described above,5.1.1 with the analysis sets stated in Section 5. Same analysis will be performed for SAS as well.

## 5.2. Secondary Endpoints

#### 5.2.1. GC IL-2

GC IL-2 change from pre GC to post GC at Day 15 will be analyzed.

#### 5.2.1.1. Main Analysis

Log transformed GC IL-2 change from pre GC to post GC at Day 15 will be analyzed using ANCOVA model as described in Section 4.2.1 based on Estimand 2 (see Section 1.1.2) for the BS. The LSM change (log transformed), LSM difference of LSM change (log transformed) between KAN-101 and PBO, 95% CI, and p-value will be presented. Exponentially transformed values for LSM, LSM difference, 95% CI will be presented as well.

#### 5.2.1.2. Sensitivity/Supplementary Analysis

The above analysis will also be performed for the log transformed GC IL-2 for the analysis sets stated in Section 5 as a supplementary analysis.

#### 5.2.2. IEL density in duodenum biopsy

Summary statistics will be provided for observed values for IEL and the change from baseline at Day 29.

#### 5.2.2.1. Main Analysis

IEL change from baseline at Day 29 will be analyzed using ANCOVA model as described in Section 4.2.1 based on Estimand 3 (see Section 1.1.2) for the FAS. The LSM change, LSM difference of LSM change between KAN-101 and PBO, 95% CI, and p-value will be presented.

#### 5.2.2. Sensitivity/Supplementary Analysis

The above analysis will be performed for PPS and the SAS as a sensitivity/supplementary analyses.

#### 5.2.3. Incidence and Severity of TEAEs as Assessed by the CTCAE

See safety Section 5.5.1.

#### 5.2.4. Incidence of Development of ADA During the Study

Participants positive for ADA (screening, confirmatory, specificity and titer) will be summarized by treatment group and timepoint with number and percent for the SAS.

#### 5.2.5. PK Concentration

PK concentration will be descriptively summarized by treatment group and nominal timepoints with number of observations, mean, SD, min, 1<sup>st</sup>, 2<sup>nd</sup> and 3<sup>rd</sup> quartiles, max for PKAS. Line plot will be provided by treatment group for mean (+/-SD) concentration-time profiles using linear and semi-log scale

#### 5.2.6. PK Parameters

PK parameters listed in Section 2.2 (AUC<sub>inf</sub>, AUC<sub>last</sub>,  $C_{max}$ ,  $T_{max}$ , and  $t_{1/2}$ ) will be descriptively summarized by treatment group with number of observations, mean, SD, min,  $1^{st}$ ,  $2^{nd}$  and  $3^{rd}$  quartiles, max, GM, and %CV for PKAS. No GM and %CV for  $T_{max}$ .

#### 5.3. Tertiary/Exploratory

#### 5.3.1. Change from baseline in Marsh-Oberhuber score at Day 29

Marsh-Oberhuber score at baseline and Day 29 observed values will be summarized with number of observations, frequency and percentage for each category. The shift from baseline to Day 29 will be summarized as well. The analysis sets used for this endpoint is found in Section 5.

#### 5.3.2. CDSD

The weekly average score of each severity item and frequency question of CDSD (Diarrhea, Abdominal Pain, Bloating, Nausea, Number of times Vomiting, Tiredness, Number of Bowel Movements and Number of events of Diarrhea) as well as the weekly average CDSD Total Score, weekly average CDSD GI Domain Score (see Section 2.3 and Appendix 2.2) and change from baseline will be descriptively summarized as stated in Secton 5 for each treatment group by timepoint.

The change from baseline for weekly average of each of the 5 severity items and 3 frequency questions, the weekly average CDSD Total Score, and the weekly average CDSD GI Domain Score will be analyzed using ANCOVA models in Section 4.2.1 by timepoint. LSM of the treatments with 95% CI, LSM of the treatment difference with PBO, p-value and 95% CI will be generated.

If there are multiple records on a same day, the earliest one will be used for analysis.

The analysis set(s) used for these endpoints are found in Section 5.

#### **Weekly Time Definitions:**

| | Regardless the day of Day 15 GC | Day 15 GC is at day 14 | Day 15 GC is at day 15 | Day 15 GC is at day 16 | Day 15 GC is at day 17 |
|---|---|---|---|---|---|
| Baseline | Day -7 to -1 | | | | |
| Week 1 | Day 1 to 7 | | | | |
| Week 2 | | Day 8 to 13 | Day 8 to 14 | Day 8 to 15 | Day 8 to 16 |
| Week 3 | | Day 14 to 21 | Day 15 to 21 | Day 16 to 21 | Day 17 to 21 |
| Week 4 | Day 22 to 28 | | | | |
| Week 5 | Day 29 to 35 | | | | |
| Week 6 | Day 36 to 42 | | | | |

In addition, the change from baseline in CDSD Nausea score and vomiting frequency for Day 15, 3-day average and 7-day average (weekly average) score, will be summarized as stated above, and analyzed within placebo and KAN treatment, evaluating the paired difference from baseline using the Wilcoxon Signed-rank test. The Mann-Whitney U test (Wilcoxon Rank Sum test) will be used to test the difference in the change from baseline for placebo vs KAN-101. The median difference between treatment groups estimated by the Hodges–Lehmann method along with the 95% CI will be reported as well.

Line plots by treatment group will be provided for LSM 95% CI).

#### 5.3.2.1. PGIS

PGIS and change from baseline will be descriptively summarized as stated in Section 5. The change from baseline will be analyzed using ANCOVA models in Section 4.2.1 by timepoint. LSM of the treatments, LSM of the treatment difference with PBO, p-value and 95% CI will be generated.

The analysis will be performed for all collected data as stated in Section 5.

#### 5.3.2.2. PGIC

PGIC will be descriptively summarized as stated in Section 5.

The analysis will be performed for all collected data as stated in Section 5.

#### 5.3.2.3. Subset Analyses

N/A

#### 5.4. Baseline and Other Summaries and Analyses

#### 5.4.1. Baseline Summaries

Demographic and baseline characteristics listed in Section 2.4 will be summarized according to Sponsor's reporting standards for the SAS.

#### 5.4.2. Study Conduct and Subject Disposition

Participants evaluation, disposition, discontinuation will be summarized for the SAS according to Sponsor's reporting standards.

#### 5.4.3. Study Treatment Exposure

The exposure to study drug will be summarized by treatment group for number of doses of study intervention applied for the SAS.

#### 5.4.4. Gluten Challenge

GC will be summarized by number and percentage of participants completed number of days of GC for the SAS, FAS, and PPS. GC can be mixed with liquid such as water, lactose-free mild or lactose-free chocolate milk, fruit juice (no prune, pear, or apricot), sports drink. The number and percentage of participants with mixture to GC will be summarized by treatment, mixture type, and GC day for the SAS, FAS, and PPS

#### 5.4.5. Concomitant Medications and Non-Drug Treatments

Prior drug and non-drug treatment, concomitant drug and non-drug treatment will be summarized according to Sponsor's reporting standards.

#### 5.5. Safety Summaries and Analyses

Safety analyses will be based on the SAS.

All clinical TEAEs, SAEs, withdrawal due to AEs, vital signs and safety laboratory data will be reviewed on an ongoing basis during the study to evaluate the safety of participants.

Safety data will be presented in tabular and/or graphical format and summarized descriptively, where appropriate. All safety endpoints will be listed and summarized in accordance with Sponsor's Standards. Categorical outcomes (eg, AEs) will be summarized by participant counts and percentage. Continuous outcome will be summarized using N, mean, median, SD, min, max. Participant listings will be produced for these safety endpoints accordingly.

#### 5.5.1. Adverse Events

Adverse events will be summarized for the SAS according to Sponsor's reporting standards for

- TEAEs
- Serious AEs (SAEs)
- TEAEs will be summarized by the number of participants reporting any TEAE, system organ class (SOC), preferred term (PT), severity, relationship to investigational product (based on investigator's judgement).
- CTCAE is used to grade the severity of AEs. TEAEs related to GC and infusion-related reactions (IRR) will also be summarized separately.
- SAEs will be summarized by SOC and PT, and individual SAEs will be listed by participant.

A list of subjects who prematurely discontinue from the study due to an AE will be provided as well.

#### 5.5.2. Safety Laboratory Data

Clinical safety laboratory values listed in Section 2.5.2 and change from baseline and clinically significant change will be summarized according to Sponsor's standards.

#### 5.5.3. Vital Signs

Vital signs and change from baseline and clinically significant change will be summarized according to Sponsor's standards.

#### 6. INTERIM ANALYSES

An interim analysis (IA) will be conducted to assess efficacy and safety after approximately 13 participants from each group have completed through the Day 29 visit including histology assessments.

Before any interim analysis is performed, the details of the objectives, decision criteria, dissemination plan, and method of maintaining the study blind (if applicable) as per the sponsor's or sponsor designee's SOPs will be documented in the Interim Analysis Plan.

#### 7. CHANGES FROM PROTOCOL

- Sample size calculation was updated to include consideration for multiple looks. Decision rules were also updated.
- Sensitivity/Supplementary analyses were updated with the new populations.

- Prohibited medications are considered in the study set definitions with the other intercurrent events (noncompliance with study medications and noncompliance with gluten challenge).
- An additional study set was added for IL2 called the BAS.

#### 8. REFERENCES

1. Protocol KAN-101-03 Amendment 1 20March2024.

# **APPENDICES**

# Appendix 1. Summary of Efficacy/Exploratory Analyses

| Endpoint | Analysis Type | Population | Analysis Model |
|---|---|---|---|
| Change from<br>baseline in Vh:Cd<br>ratio at Day 29 | Summary | FAS | N/A |
| | Main analysis | FAS | ANCOVA with terms treatment, baseline |
| | Sensitivity/supplementary analysis | PPS, SAS | ANCOVA with terms treatment, baseline |
| GC IL-2 (log-<br>transformed) change<br>from Day 15 pre-GC<br>to Day 15 post GC | Summary | BAS | N/A |
| | Analysis | BAS | ANCOVA with terms treatment, baseline |
| | Sensitivity/supplementary analysis | PPS, SAS | ANCOVA with terms treatment, baseline |
| Changes from<br>baseline in IEL<br>density in duodenum<br>biopsy after 2-week<br>GC (at Day 29) | Summary | FAS | N/A |
| | Analysis | FAS | ANCOVA with terms treatment, baseline |
| | Sensitivity/supplementary analysis | PPS, SAS | ANCOVA with terms treatment, baseline |

| Endpoint | Analysis Type | Population | <b>Analysis Model</b> |
|---|---|---|---|
| CDSD change from baseline at each timepoint | Summary | FAS | N/A |
| | Analysis | FAS | ANCOVA with terms treatment, baseline |
| | Sensitivity/supplementary analysis | PPS, SAS | ANCOVA with terms treatment, baseline |
| CDSD 1-Day, 3-Day, 7-Day Nausea Score and Vomiting Frequency and change from baseline at each timepoint postgluten challenge | Summary | FAS | Observed cases |
| | Analysis | FAS | All data collected will be included regardless of intercurrent events. Missing data will not be imputed. Wilcoxon Signedrank test for change from baseline within each group |
| | Analysis | FAS | All data collected will be included regardless of intercurrent events. Missing data will not be imputed. Mann-Whitney U test (Wilcoxon |

| Endpoint | Analysis Type | Population | Analysis Model |
|---|---|---|---|
| | | | Rank Sum test) for<br>comparison of<br>placebo vs KAN<br>group for change<br>from baseline |
| PGIS change from baseline at each timepoint | Summary | FAS | N/A |
| | Analysis | FAS | ANCOVA with terms treatment, baseline |
| PGIC at each timepoint | Summary | FAS | N/A |
| | Analysis | FAS | ANOVA with term treatment |
| Marsh- Oberhuber score | Summary | FAS, PPS,<br>SAS | N/A |

#### **Appendix 2. Data Derivation Details**

#### Appendix 2.1. Definition and Use of Analysis Windows in Reporting

Analysis windows will be used for PROs and vital signs, and laboratory tests.

If more than one observation from the same participant falls into the same analysis window, the value closest to the targeted day will be used as the observation for that visit. All observations will, however, be included in the listings.

Table 3 Analysis Windows for PGIS and PGIC

| Visit Label | Targeted Day | Analysis window for data sets |
|---|---|---|
| Baseline (Screening up to | Day 1 | Last observation up to and including first |
| first dosing date) | - | dosing date |
| Day 15 | Day 15 | After last dose – First day of GC |
| Day 29 | Day 29 | Second day of GC – Day 35 |
| Day 42 | Day 42 | Day 36 – end of study |

**Table 4 Analysis Windows for Vital Signs** 

| Visit Label | Targeted Day | Analysis window for data sets |
|---|---|---|
| Baseline (Screening up to first dosing date) | Day 1 | Last observation up to first dosing |
| Day 1 during dosing | Day 1 during dosing | Start of Day 1 dosing to end of Day 1 dosing |
| Day 1 after dosing | Day 1 after dosing | End of Day 1 dosing to end of Day 1 |
| Day 4 before dosing | Day 4 pre-dosing | Day 2 - Day 4 pre-dosing |
| Day 4 during dosing | Day 4 during dosing | Day 4 start of dosing - Day 4 end of dosing |
| Day 4 after dosing | Day 4 after dosing | Day 4 end of dosing - end of Day 4 |
| Day 7 before dosing | Day 7 pre-dosing | Day 5 - Day 7 pre-dosing |
| Day 7 during dosing | Day 7 pre-dosing | Day 7 start of dosing - Day 7 end of dosing |
| Day 7 after dosing | Day 7 after dosing | Day 7 end of dosing - end of Day 7 |
| Day 15 | Day 15 pre-GC | Day 8 - pre-GC of first GC day |
| Day 29 | Day 29 | After GC of first GC day – Day 35 |
| Day 42 | Day 42 | Day 36 – end of study |

#### **Table 5 Analysis Windows for Laboratory Tests**

| Visit Label | Targeted Day | Analysis window for data sets |
|---|---|---|
| Baseline (Screening up to | Day 1 | Last observation up to first dosing |
| first dosing date) | | |
| Day 4 | Day 4 pre-dosing | Day 1 after dosing - Day 4 pre-dosing |
| Day 7 | Day 7 pre-dosing | Day 4 after dosing - Day 7 pre-dosing |
| Day 15 | Day 15 pre-GC | Day 7 after dosing - pre-GC of first GC |
| | | day |
| Day 29 | Day 29 | post-GC of first GC day – Day 35 |
| Day 42 | Day 42 | Day 36 – end of study |

## **Table 6 Analysis Windows for ADA**

| Visit Label | Targeted Day | Analysis window for data sets |
|---|---|---|
| Baseline (Screening up to | Day 1 pre-dosing | Last observation prior to first |
| first dosing) | | dosing date |
| Day 7 | Day 7 pre-dosing | Day 2 - Day 7 pre-dosing |
| Day 29 | Day 29 | Day 8 – Day 35 |
| Day 42 | Day 42 | Day 36 – end of study |

# Table 7 Analysis Windows for biopsy endpoints (Vh:Cd ratio, IEL density, Marsh-Oberhuber score)

| Visit Label | Targeted Day | Analysis window for data sets |
|---|---|---|
| Baseline (Screening up to | Day 1 pre-dosing | Last observation prior to first |
| first dosing) | | dosing date |
| Day 29 | Day 29 | Day 22 – Day 43 |

#### Table 8 Analysis Windows for IL-2 and CDSD at Day 15 (first GC Day)

| Visit Label | Targeted Day | Analysis window for data sets |
|-------------|--------------|--------------------------------|
| Day 15 | Day 15 | The first GC day, Day 14 – Day |
| | | 17 |

Appendix 2.2. Celiac Disease Symptom Diary (CDSD)



**Appendix 2.3. Patient Global Impression of Severity (PGIS)** 



**Appendix 2.4. Patient Global Impression of Change (PGIC)** 



# **Appendix 3. List of Abbreviations**

| the time of the last quantifiable concentration (C <sub>last</sub> ) BAS Biomarker analysis set BP blood pressure CDSD celiac disease symptom diary CeD celiac disease CI Confidence interval C <sub>max</sub> maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | Abbreviation | Term |
|---|---|---|
| AE adverse event ALT alanine aminotransferase ANCOVA analysis of covariance ANOVA Analysis of variance AST aspartate aminotransferase AUCinf area under the plasma-concentration curve from time 0 extrapolated to infinite time AUClast area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (Clast) BAS Biomarker analysis set BP blood pressure CDSD celiac disease symptom diary CeD celiac disease CI Confidence interval Cmax maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-friee diet GI Gastrointestinal GM geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | ADA | anti-drug antibodies |
| ALT alanine aminotransferase ANCOVA analysis of covariance ANOVA Analysis of variance AST aspartate aminotransferase AUC <sub>inf</sub> area under the plasma-concentration curve from time 0 extrapolated to infinite time AUC <sub>last</sub> area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (C <sub>last</sub> ) BAS Biomarker analysis set BP blood pressure CDSD celiac disease symptom diary CeD celiac disease CI Confidence interval Cmax maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GMM geometric mean GMR geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | ADL | activity/activities of daily living |
| ANCOVA Analysis of covariance ANOVA Analysis of variance AST aspartate aminotransferase AUC <sub>inf</sub> area under the plasma-concentration curve from time 0 extrapolated to infinite time AUC <sub>last</sub> area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (C <sub>last</sub> ) BAS Biomarker analysis set BP blood pressure CDSD celiac disease symptom diary CeD celiac disease CI Confidence interval Cmax maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten-challenge GFD gluten-free diet GI GGA Gastrointestinal GM geometric mean GMR geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max min minimum N/A not applicable PBO PGIC Patient Global Impression of Change | AE | adverse event |
| ANOVA Analysis of variance AST aspartate aminotransferase AUC <sub>inf</sub> area under the plasma-concentration curve from time 0 extrapolated to infinite time AUC <sub>last</sub> area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (C <sub>last</sub> ) BAS Biomarker analysis set BP blood pressure CDSD celiac disease symptom diary CeD celiac disease CI Confidence interval Cmax maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | ALT | alanine aminotransferase |
| AST aspartate aminotransferase AUC <sub>inf</sub> area under the plasma-concentration curve from time 0 extrapolated to infinite time AUC <sub>last</sub> area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (C <sub>last</sub> ) BAS Biomarker analysis set BP blood pressure CDSD celiac disease symptom diary CeD celiac disease CI Confidence interval C <sub>max</sub> maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | ANCOVA | analysis of covariance |
| AUC <sub>inf</sub> area under the plasma-concentration curve from time 0 extrapolated to infinite time AUC <sub>inst</sub> area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (C <sub>last</sub> ) BAS Biomarker analysis set BP blood pressure CDSD celiac disease symptom diary CeD celiac disease CI Confidence interval C <sub>max</sub> maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | ANOVA | Analysis of variance |
| extrapolated to infinite time AUC <sub>last</sub> area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (C <sub>last</sub> ) BAS Biomarker analysis set BP blood pressure CDSD celiac disease symptom diary CeD celiac disease CI Confidence interval Cmax maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min min minimum N/A not applicable PBO PGIC Patient Global Impression of Change | AST | aspartate aminotransferase |
| AUC <sub>last</sub> area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (C <sub>last</sub> ) BAS Biomarker analysis set BP blood pressure CDSD celiac disease CI Confidence interval C <sub>max</sub> maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO PGIC Patient Global Impression of Change | AUCinf | area under the plasma-concentration curve from time 0 |
| the time of the last quantifiable concentration (C <sub>last</sub> ) BAS Biomarker analysis set BP blood pressure CDSD celiac disease symptom diary CeD celiac disease CI Confidence interval Cmax maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | | |
| BAS Biomarker analysis set BP blood pressure CDSD celiac disease symptom diary CeD celiac disease CI Confidence interval Cmax maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | AUC <sub>last</sub> | |
| BP blood pressure CDSD celiac disease symptom diary CeD celiac disease CI Confidence interval Cmax maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GMM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO Patient Global Impression of Change | | |
| CDSD celiac disease symptom diary CeD celiac disease CI Confidence interval Cmax maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO PGIC Patient Global Impression of Change | | · |
| CeD celiac disease CI Confidence interval Cmax maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO Patient Global Impression of Change | | - |
| CI Confidence interval Cmax maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO Patient Global Impression of Change | | |
| Cmax maximum observed concentration CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | | |
| CTCAE common terminology criteria for adverse events CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | | |
| CV coefficient of variation DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | $C_{max}$ | |
| DSMB data safety monitoring board ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | | |
| ET early termination FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | CV | coefficient of variation |
| FAS full analysis set GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | DSMB | data safety monitoring board |
| GC gluten challenge GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | ET | early termination |
| GFD gluten-free diet GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | FAS | full analysis set |
| GI Gastrointestinal GM geometric mean GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | GC | gluten challenge |
| GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | GFD | gluten-free diet |
| GMR geometric mean ratio ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | GI | Gastrointestinal |
| ICD informed consent document IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | GM | geometric mean |
| IL-2 interleukin-2 IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | GMR | geometric mean ratio |
| IRR infusion-related reactions LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | ICD | informed consent document |
| LLOQ Lower Limit of Quantification max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | IL-2 | interleukin-2 |
| max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | IRR | infusion-related reactions |
| max maximum min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | | |
| min minimum N/A not applicable PBO placebo PGIC Patient Global Impression of Change | LLOQ | Lower Limit of Quantification |
| N/A not applicable PBO placebo PGIC Patient Global Impression of Change | max | maximum |
| PBO placebo PGIC Patient Global Impression of Change | min | minimum |
| PGIC Patient Global Impression of Change | N/A | not applicable |
| 1 C | PBO | |
| | PGIC | Patient Global Impression of Change |
| | PGIS | |

| Abbreviation | Term |
|------------------|-----------------------------------|
| PK | pharmacokinetic(s) |
| PKAS | PK analysis set |
| PRO | patient-reported outcome |
| PT | preferred term |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SAS | Safety analysis set |
| SD | standard deviation |
| SOC | system organ class |
| t <sub>1/2</sub> | terminal phase half-life |
| TEAE | treatment -emergent adverse event |
| $T_{\text{max}}$ | time to reach C <sub>max</sub> |
| ULN | upper limit of normal |